CLINICAL TRIAL: NCT02837549
Title: Novel Rehabilitation Strategies to Improve Arm Function in Patients With Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Susan Murphy, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00117117
Record Dates: First submitted 2016-07-05; First posted 2016-07-19 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Scleroderma; Ssc
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Occupational therapy treatment (Experimental): Participants will undergo the following as appropriate:
  1. Thermal Modalities Hot packs, focused on areas with limitations Paraffin, focused on digital limitations
  2. Application of the Physiotouch (a low-intensity negative pressure device)
  3. Passive Range of Motion
  4. Active Range of Motion
  5. Functional Activities
  Interventions: Other: Occupational therapy treatment

INTERVENTIONS:
Other: Occupational therapy treatment — This intervention includes various thermal modalities, manual therapy, Physiotouch (Healthy Life Devices Ltd) and education
  Other Names: Upper Extremity Rehabilitation

SUMMARY:
The purpose of this study is to determine the feasibility and preliminary effects of a novel treatment approach to improve arm function in patients with scleroderma who have upper extremity contractures. It is a Phase 1, one arm trial in which participants will be assessed at baseline, 4 weeks, and 8 weeks. The rehabilitation intervention will involve 8 individual sessions with an occupational therapist. Feasibility of the procedures is a major focus of this project.

DETAILED DESCRIPTION:
Our specific aims are to:

1. Determine the feasibility of a novel rehabilitation strategy provided at the University of Michigan Scleroderma Clinic to scleroderma patients who have upper extremity contractures.

   Investigators will assess 3 main aspects of the process that are key to the success of a larger study including the proportion of eligible people who enroll in the study, rate of adherence to the treatment protocol, and the time it takes to conduct sessions including treatment and outcome assessment completion. Based on a framework of recommendations for well-designed pilot studies [1], investigators have set the following criteria for success to examine these aspects:
   1. At least 50% of participants who are eligible for the study will enroll.
   2. At least 80% of participants will attend all treatment sessions.
   3. The 3 sessions involving both treatment and outcome assessments will not last on average more than 2 hours.
2. Develop a standardized treatment manual to train therapists to provide this treatment to their patients.

   A standardized treatment manual for therapists is a critical component needed to ensure consistency in a larger multi-site trial. This manual will be drafted for use in this study and refined as needed.
3. Establish preliminary effects of this 8-week rehabilitation program on improving arm function.

Investigators hypothesize that participants with scleroderma will have significant improvements in the QuickDASH disability measure at post test. Although the investigators think large effects will be shown, this study will allow us to determine estimates of the effects and the variability for power calculations in a multi-site trial.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of scleroderma (localized or generalized morphea)
* Have a contracture of the hand and other joint in at least one arm, such as wrist, elbow, or shoulder, with the ability to demonstrate active range of motion in that arm
* Willing to travel to participate in therapy and outcome assessments.
* English speaking

Exclusion Criteria:

* active hand ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
quickDASH | change over 8 weeks
  self-report questionnaire of physical function and symptoms

SECONDARY OUTCOMES:
Upper extremity range of motion | change over 8 weeks
  Active and Passive Range of Motion measured by goniometer
Coordination | change over 8 weeks
  9 hole peg test
Grip Strength | change over 8 weeks
  dynanometer
Physical Function | change over 8 weeks
  PROMIS physical function 8-item short form

CONTACTS AND LOCATIONS:
Overall Officials: Susan Murphy, ScD, Principal Investigator — University of Michigan - Department of Physical Medicine and Rehabilitation
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
upon written request

REFERENCES:
- [Derived] Murphy SL, Barber MW, Homer K, Dodge C, Cutter GR, Khanna D. Occupational Therapy Treatment to Improve Upper Extremity Function in Individuals with Early Systemic Sclerosis: A Pilot Study. Arthritis Care Res (Hoboken). 2018 Nov;70(11):1653-1660. doi: 10.1002/acr.23522. PMID 29381834